CLINICAL TRIAL: NCT03442517
Title: Learning About Techniques to Create Healthy Infants Through Nutrition and Proper Growth
Brief Title: The LATCHING Pilot Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00140506
Record Dates: First submitted 2017-12-20; First posted 2018-02-22 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Breastfeeding
Keywords: group-based counseling; phone counseling; conference calls
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-based phone counseling (GBPC) (Experimental): Participants will take part in weekly group-based phone counseling sessions for 6 weeks starting between 16-30 weeks of pregnancy.
  Interventions: Behavioral: Behavior Lifestyle Intervention
- Usual prenatal care (Active Comparator): Participants will continue their usual prenatal care.
  Interventions: Other: Usual prenatal care

INTERVENTIONS:
Behavioral: Behavior Lifestyle Intervention — Participants will be involved in group-based counseling. Sessions will be about 1 hour each and comprise up to 10 people. The sessions will be led by a trained health educator. The calls will be a chance for participants to discuss challenges with breastfeeding, problem solving skills, educational information, and discuss balanced diet topics.
  Other Names: Group-based phone counseling
  Arms: Group-based phone counseling (GBPC)
Other: Usual prenatal care — Participants will receive the standard education given by their OBGYN or other healthcare provider. No additional breastfeeding, nutrition or postpartum weight loss education will be provided to participants by the investigators during pregnancy. After delivery, participants will follow normal pediatric visit schedule.
  Arms: Usual prenatal care

SUMMARY:
The purpose of this study is to learn if group-based phone counseling is effective for increasing breastfeeding rates, reducing the early introduction of solids and increasing maternal weight loss after pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women who are 9-30 weeks in gestation that have not previously met breastfeeding recommendations
* Speak and understand English

Exclusion Criteria:

* Women with pregnancies conceived using fertility treatments, those at high risk for pre-term delivery, those with multiple gestation (ie. twins, triplets, etc), or pregnancies complicated by morbid obesity (BMI>40), diabetes (pre-gestational or gestational), hypertension, metabolic dysfunction, etc.
* Women who have previously exclusively breastfed an infant for three or more months

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2017-04-29 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Differences in infant feeding progression | Month 6
Proportion of women exclusively breastfeeding | Month 6
Proportion of women who introduce solids | Month 4

SECONDARY OUTCOMES:
Subject satisfaction and acceptability of intervention | Week 24
  Structured interviews will be used to determine subject satisfaction. Structured interviews will obtain descriptive data regarding problems encountered by participants during the intervention, areas of intervention strength and weakness, information participants found helpful and information participants wish they had been given during the intervention, and ways the overall intervention could be improved.
Intervention compliance | Week 24
  Compliance rates will be calculated from participants that attend at least 66.6% (at least 4 sessions) of GBPC sessions.
Study Retention | Month 6
  Retention rates will be calculated from participants who complete feeding questionnaire data at 6 months.

OTHER OUTCOMES:
Differences in infant feeding progression | Week 2
Differences in infant feeding progression | Month 2
Differences in infant feeding progression | Month 4

CONTACTS AND LOCATIONS:
Overall Officials: Holly Hull, PhD, Principal Investigator — University of Kansas Medical Center
Locations (3):
- United States (3):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Priority Care Pediatrics, LLC, Kansas City, Missouri
  - Northland Obstetrics & Gynecology, Inc., Liberty, Missouri

REFERENCES:
- [Derived] Cauble JS, Herman A, Wick J, Goetz J, Daley CM, Sullivan DK, Hull HR. A prenatal group based phone counseling intervention to improve breastfeeding rates and complementary feeding: a randomized, controlled pilot and feasibility trial. BMC Pregnancy Childbirth. 2021 Jul 22;21(1):521. doi: 10.1186/s12884-021-03976-2. PMID 34294051